CLINICAL TRIAL: NCT05937633
Title: A Study to Evaluate the Effect of Transformational Leadership Programme on Unit Charge Nurses Leadership Practices in Hamad Medical Corporation: A Randomized Controlled Trial
Brief Title: Effect of Transformational Leadership Programme on Unit Charge Nurses Leadership Practices
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: MRC-01-22-386
Record Dates: First submitted 2023-06-06; First posted 2023-07-10 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2022-08

CONDITIONS: Leadership

STUDY DESIGN:
Intervention Model Description: This study uses a prospective, parallel group, randomized control group design to compare those received transformational leadership programme to standard educational booklet among charge nurses.
  The samples will be divided into experimental and control group by randomly assigning the subjects to each group.
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the study the subjects and investigator are not masked. However the outcome assessors are marked for analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tranformational Education (Experimental): A total of 82 Participants will be assigned to experimental group. Transformational educational programme is administered to all the participants.
  Interventions: Other: Transformational Education Programme
- Educational Booklet (No Intervention): Study participants (Charge Nurses and Acting Charge Nurses) of educational booklet group will be distributed with educational booklet.

INTERVENTIONS:
Other: Transformational Education Programme — An evidence based targeted transformational leadership programme is designed to provide charge nurses an opportunity to develop transformational leadership knowledge and skill.
  The programme includes a 2-day activity based educational training. A prereading booklet will be given prior to the educational activity aimed at enhancing the engagement of the participants. The educational programme comprises of the following contents: Concept of leadership and work engagement, transactional and transformational leadership styles, advantages, and disadvantages of transformational leaders. qualities of transformational leaders, 5- Practices of exemplary leadership practice, the 10 commitments of transformational leadership and developing transformational leadership skills.
  Arms: Tranformational Education

SUMMARY:
Nurse leaders need to be visionary adapting to the fast-paced environments and influence their followers in achievement of the goals. Transformational leadership is one of the most widely used style of leadership across the disciplines. Transformational leadership has been shown to enhance nurse satisfaction, recruitment, and retention to promote healthy environment. The aim of this study is to assess the impact of an educational programme on the transformational leadership characteristics of charge nurses and their relationship to nurse's work engagement. An interactive transformational leadership programme targeting specific leadership knowledge and skills will be administered and evaluated.

DETAILED DESCRIPTION:
Leadership is defined as a process that persons usually perform to bring forth the best from themselves and their followers. After extensive review of literature it is identified that there is dearth of studies on the use of leadership programme among charge nurses. Most of the studies conducted on the leadership styles and their characteristics are correlational in nature where the causality is not measured.

It is identified that there were few studies conducted on leadership styles in Qatar, but the investigators did not find studies conducted on effectiveness of targeted transformational leadership development interventions among charge nurses. The investigator is interested in developing a targeted leadership development programme based on transformational leadership theory and strong evidence to implement among charge nurses.

Based on the current health scenario and considering the challenges posed by Covid-19, there is a need to develop transformational leadership skills of charge nurses with a view to develop future leaders. In this context the investigator is interested to conduct a study to answer the question, does targeted Transformational Leadership Programme change Transformational leadership practices among charge nurses?

The aim of the study is to evaluate the effect of transformational leadership programme on unit charge nurses leadership practices. This study uses a prospective, parallel group, randomized control group design to compare those received transformational leadership programme to standard educational booklet among charge nurses.The samples will be divided into two groups and subjects will be randomly assigned to both groups.The research team will use blocked randomization method for randomly assigning the subjects to both arms.The study also explores the relationship between transformational leadership practices and work engagement among unit charge nurses.

A total of 164 samples are needed for the study. The samples will be randomly assigned to the two arms. The leadership practice inventory will be used for assessment of leadership practices of charge nurses. This tool is considered as valid and reliable. Assessment using Leadership Practice Inventory will be done at the beginning of administering the intervention and after 3 months of training. Work engagement of staff nurses will be assessed using Utrecht Work Engagement Scale.

An evidence based targeted transformational leadership programme is designed by the research team and validated. The programme includes a 2-day activity based educational training. Pre Reading material will be sent to study participants prior to the educational activity. The educational programme comprises of the following contents: Concept of leadership and work engagement, transactional and transformational leadership styles, advantages and disadvantages of transformational leaders. qualities of transformational leaders, 5- Practices of exemplary leadership practice, the 10 commitments of transformational leadership and developing transformational leadership skills for nurses.

This educational programme will be administered to transformational leadership training group. Based on the feedback obtained from participants reflective assignments will be planned and evaluated. The participants are encouraged to put into practice the knowledge and skills gained during the educational programme.

The subjects from control group will receive a educational booklet for self reading. The same leadership practice inventory will be used for assessment of leadership practices of subjects from the educational booklet group.

ELIGIBILITY:
Inclusion Criteria:

* Working as a Charge Nurse or Acting Charge Nurse with all responsibilities of the nursing unit.
* Consent to participate from the Nursing Administration. (Executive Director of Nursing and respective Directors of Nursing)
* Anticipated availability for the complete programme.

Exclusion Criteria:

* Charge Nurses or Acting Charge Nurses who are currently undergoing any Leadership Training Programme.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in transformational leadership behavior of charge nurses. | 3 Months
  The primary target outcome is anticipated change in transformational leadership behavior of charge nurses assessed by using Leadership Practice Inventory. Leadership practice inventory is a standardized tool to assess the transformational leadership practices which is valid and reliable.
  The Inventory examines five basic leadership practices: modeling the way, inspiring a shared vision, challenging the process, enabling others to act, encouraging the heart. Each of these leadership practices are measured by six items rated by 10 Point Likert Scale (1= almost never, 10= almost always). Each sub-scale ranges from 6 to 60, with higher scores indicating better transformational practices.
  The research team are expecting a change in the transformational leadership practice of the charge nurses from the transformational educational training group as compared with standard educational booklet group.

SECONDARY OUTCOMES:
Change in work engagement of staff nurses. | 3 Months
  The study also aims to assess the work engagement of staff nurses using Utrecht Work Engagement Scale. The Utrecht Work Engagement Scale is a valid tool that includes 3 dimensions of work engagement: vigor (6 items), absorption (6 items), and dedication (5 items).
  A 7-point Likert scale is used, with scores ranging from 0 (never) to 6 (always); higher scores indicate higher levels of engagement.
  The researchers are anticipating a correlation between the transformational leadership practices of charge nurses to have an impact on their sub ordinates work engagement. Hence work engagement of staff nurses will be measured using the Utrecht work engagement scale.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Wesley Devanesan, Masters, Principal Investigator — Al Wakra Hospital
Locations (1):
- Hamad Medical Corporation, Doha, Qatar

IPD SHARING:
Plan to Share IPD: No
Post data collection, all the data will be stored in a data base by the principal investigator. Only PI will have access to the data base with a password. The Data will be shared only with the concerned research team member. The data will be stored at Nursing Supervisor Department at Al- Wakra Hospital.
  Subject identifiers will not be shared outside HMC.